CLINICAL TRIAL: NCT00761462
Title: A Prospective, Open-label, Non-randomized, Naturalistic, Long-term Safety Surveillance, Observational Study of Either Ciprofloxacin (Either as Oral Suspension, Oral Tablets or Sequential IV Followed by Oral Therapy or Purely IV Therapy) or a Non-quinolone Antibiotic (Either as Oral Suspension, Oral Tablets or Sequential IV Followed by Oral Therapy or Purely IV Therapy) in the Treatment of Pediatric Patients With Infectious Diagnoses
Brief Title: BAY 0 9867 Cipro Pediatric Use Study (QUIP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100201; 2014-004622-18 (EudraCT Number)
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Results first posted 2009-04-14 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Infectious Diseases
Keywords: Pediatrics; Safety; Musculoskeletal System; Neurologic Manifestations; Joint Diseases; Joint Deformities, Acquired
MeSH Terms: conditions — Communicable Diseases; Neurologic Manifestations; Joint Diseases; Joint Deformities, Acquired | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ciprofloxacin (Experimental): Subjects receiving Ciprofloxacin (group followed-up for 5 years)
  Interventions: Drug: Ciprofloxacin
- Non-quinolone antibiotic (Active Comparator): Subjects receiving non-quinolone antibiotic (group followed-up for 2 years)
  Interventions: Drug: Non-quinolone antibiotic

INTERVENTIONS:
Drug: Ciprofloxacin — Either as oral suspension, oral tablets or sequential intravenous (IV) - oral therapy or purely IV therapy according to label
  Arms: Ciprofloxacin
Drug: Non-quinolone antibiotic — Common used dose and route
  Arms: Non-quinolone antibiotic

SUMMARY:
Objective and subjective musculoskeletal evaluations will be performed to determine differences in the ciprofloxacin versus non-quinolone treated pediatric patients so that we can tell what the natural occurrence of such musculoskeletal conditions is in the general pediatric population.

DETAILED DESCRIPTION:
This study is classified as "interventional" due to study-specific medical examinations and interventions. Regarding the study drug intake, routine administration is observed only, there is no intervention in study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >/= 2 months of age through 16 years of age
* A parent/caregiver must sign an informed consent
* Patient must provide assent, as appropriate based on local institutional review board guidelines

Exclusion Criteria:

* Patients presenting with the following conditions:

  * exacerbations of cystic fibrosis (CF)
  * meningitis
  * Brain abscess
  * bacterial endocarditis,
  * Bone and joint infections
* having any of the following conditions but lacking a personal history may be admitted to the trial:

  * Arthritis
  * Juvenile rheumatoid arthritis (JRA)
  * Rheumatoid arthritis (RA)
  * Systemic lupus erythematosis (SLE)
  * History of rheumatic fever
  * Psoriasis
  * Inflammatory bowel disease
  * Osteoarthritis (OA)
* Known underlying rheumatological disease, joint problems known to be associated with arthropathy.
* Patients with any pre-treatment baseline musculoskeletal exam abnormalities
* Known risk of experiencing seizures, a history of any convulsive disorders
* Requiring any concomitant therapeutic course of systemic antibacterial agent
* Participation in any industry-sponsored clinical drug development study within one month prior to this study
* Known significant liver impairment (ALAT/ASAT and/or baseline bilirubin > 3 times upper limit of normal)
* Known significant renal insufficiency (calculated creatinine clearance of < 30 ml/min/1.73 m²)
* Are pregnant or lactating, or are sexually active and using unreliable contraception.

Ages: 2 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1029 (Actual)
Dates: Start 1999-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (62):
- United States (61):
  - Mobile, Alabama
  - Fort Smith, Arkansas
  - Corona, California
  - Fountain Valley, California
  - Long Beach, California
  - Orange, California
  - Pico Rivera, California
  - San Bernardino, California
  - San Luis Obispo, California
  - Centennial, Colorado
  - Denver, Colorado
  - Fort Walton Beach, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Snellville, Georgia
  - Honolulu, Hawaii
  - Idaho Falls, Idaho
  - Park Ridge, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - Bardstown, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Red Wing, Minnesota
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Hackensack, New Jersey
  - Voorhees Township, New Jersey
  - New Hyde Park, New York
  - New York, New York
  - Stony Brook, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Wilmington, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Youngstown, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Elverson, Pennsylvania
  - Havertown, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Benbrook, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Galveston, Texas
  - Houston, Texas
  - Temple, Texas
  - Layton, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Morgantown, West Virginia
- Montreal, Quebec, Canada

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Observational study in which patients were recruited between 1999 and 2002, and followed up for 5 years (ciprofloxacin patients) or 2 years (non-ciprofloxacin patients), monitoring the occurrence of musculoskeletal and central nervous system events.
Pre-assignment Details: The decision to treat with ciprofloxacin or a non-quinolone antibiotic was made prior to a patient's enrollment in the study and was based on the particular infection, type of patient, medical history, and the clinical evaluation by the prescribing physician. The study was not randomized.
Period: Treatment
Arm/Group | Ciprofloxacin | Non-quinolone Antibiotic
Started | 510 (Patients enrolled in study group) | 519 (Patients enrolled in study group)
Completed | 487 (Patients with confirmed intake of study drug) | 507 (Patients with confirmed intake of study drug)
Not Completed | 23 | 12
Not completed — Subjects never received study medication | 23 | 12
Period: 2 or 5 Years Long-term Safety Follow-up
Arm/Group | Ciprofloxacin | Non-quinolone Antibiotic
Started | 487 (Patients with confirmed intake of study drug entering long-term safety evaluation) | 507 (Patients with confirmed intake of study drug entering long-term safety evaluation)
4-6 Weeks Post Treatment | 487 | 507
1 Year Follow-up | 485 | 507
Completed | 333 (Patients under safety evaluation at end of 5 year safety Follow-up.) | 456 (Patients under safety evaluation at end of 2 year safety Follow-up.)
Not Completed | 154 | 51
Not completed — Death | 4 | 0
Not completed — Lost to Follow-up | 75 | 30
Not completed — Withdrawal by Subject | 75 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin | Non-quinolone Antibiotic | Total
Number analyzed (Participants) | 487 | 507 | 994
Age, Customized [Number; unit: participants]
  >= 2 months through 12 month | 37 | 48 | 85
  >=13 months through 23 month | 48 | 52 | 100
  >=2 years through 5 years | 150 | 165 | 315
  >= 6 years through 11 years | 194 | 223 | 417
  >=12 years through 16 years | 58 | 19 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 269 | 242 | 511
  Male | 218 | 265 | 483
Region of Enrollment [Number; unit: participants]
  United States | 476 | 503 | 979
  Canada | 11 | 4 | 15
Type of infection, pre-treatment [Number; unit: participants] — Type of infection, pre-treatment, which qualified patients for long term safety evaluation
  participants
    Category 1, Otitis Media | 143 | 207 | 350
    Category 2, Pharyngitis / Tonsillitis | 39 | 148 | 187
    Category 3, Urinary Tract | 105 | 12 | 117
    Category 4, Sinusitis | 39 | 47 | 86
    Category 5, Pyelonephritis | 24 | 8 | 32
    Category 6, Pneumonia | 12 | 17 | 29
    Category 7, Bronchitis | 7 | 7 | 14
    Category 8, Abscess | 7 | 6 | 13
    Category 9, Skin Infection | 6 | 7 | 13
    Category 10, External Otitis | 10 | 1 | 11
    Category 11, Wound Infection | 7 | 2 | 9
    Category 12, Other Respiratory Tract Infection | 2 | 6 | 8
    Category 13, Bacteremia | 6 | 1 | 7
    Category 14, Shigellosis | 7 | 0 | 7
    Category 15, Acute Bronchitis | 2 | 5 | 7
    Category 16, Pseudomonas Infections | 6 | 0 | 6
    Category 17, Abscess with cellulitis | 2 | 4 | 6
    Category 18, Mastoiditis | 5 | 0 | 5
    Category 19, Cystitis | 5 | 0 | 5
    Category 20, Other | 53 | 29 | 82

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Arthropathy (Cumulative)
Description: Arthropathy, as assessed by independent safety committee. The committee, after reviewing data related to musculoskeletal events, decided whether each patient had arthropathy or not. Each incidence includes number shown at previous time point, plus any new patients with the event. The 112/20 arthropathies are mentioned in the other Adverse Events section as well.
Time Frame: 4-6 weeks after treatment / 1 year after treatment / 2 or 5 years after treatment
Population: Patients valid for safety (all patients confirmed to have received at least one dose of study drug)
Measure: Number; unit: participants
Arm/Group | Ciprofloxacin | Non-quinolone Antibiotic
Number analyzed (Participants) | 487 | 507
participants
  4-6 weeks after treatment | 39 | 9
  1 year after treatment | 64 | 16
  2 or 5 years after treatment | 112 | 20

2. Primary Outcome: Incidence of Nervous System Events (Cumulative)
Description: Any event within the MedDRA system organ class 'Nervous System disorders'. Each incidence includes number shown at the previous time point, plus any new patients with the event.
Time Frame: 4-6 weeks after treatment / 1 year after treatment / 2 or 5 years after treatment
Population: Patients valid for safety (all patients confirmed to have received at least one dose of study drug).
Measure: Number; unit: participants
Arm/Group | Ciprofloxacin | Non-quinolone Antibiotic
Number analyzed (Participants) | 487 | 507
participants
  4-6 weeks after treatment | 38 | 10
  1 year after treatment | 49 | 13
  2 or 5 years after treatment | 56 | 17

ADVERSE EVENTS:
Arm/Group | Ciprofloxacin | Non-quinolone Antibiotic
Serious Adverse Events (participants affected / at risk) | 25/487 | 6/507
Other Adverse Events (participants affected / at risk) | 206/487 | 76/507
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciprofloxacin (N=487) | Non-quinolone Antibiotic (N=507)
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Otitis media (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Perianal abscess (Infections and infestations) | 1 | 0
Pyelonephritits (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0
Wound abscess (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Vesicoureteric reflux (Reproductive system and breast disorders) | 1 | 0
Pelvi- ureteric obstruction (Renal and urinary disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ciprofloxacin (N=487) | Non-quinolone Antibiotic (N=507)
Vomiting (Gastrointestinal disorders) | 18 | 5
Diarrhoea (Gastrointestinal disorders) | 14 | 2
Abdominal pain upper (Gastrointestinal disorders) | 12 | 5
Pyrexia (General disorders) | 19 | 7
Fatigue (General disorders) | 18 | 0
Otitis media (Infections and infestations) | 20 | 15
Upper respiratory tract infection (Infections and infestations) | 17 | 8
Joint sprain (Injury, poisoning and procedural complications) | 13 | 5
Contusion (Injury, poisoning and procedural complications) | 11 | 8
Arthropathy (Musculoskeletal and connective tissue disorders) | 112 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 84 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36 | 7
Headache (Nervous system disorders) | 31 | 8
Insomnia (Psychiatric disorders) | 17 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 3

LIMITATIONS AND CAVEATS:
The study was not randomized or blinded; the demographic and baseline infection characteristics were not comparable for the treatment groups; the long term followup times were different for the two groups (5 year versus 2 years).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less